CLINICAL TRIAL: NCT03118609
Title: Understanding the Needs of Informal Caregivers
Brief Title: Understanding Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Arlene Schmid, Prinicipal Investigator, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-6969H
Record Dates: First submitted 2017-03-20; First posted 2017-04-18 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Caregivers
Keywords: Caregivers; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: A single focus group.
  A single group will be analyzed based on survey results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers for "Understanding Needs" (Experimental): 5-8 informal caregiver participants in focus group will discuss current perceived needs.
  Up to 150 participants will complete the "Understanding Needs" survey
  Interventions: Other: Understanding Needs Survey

INTERVENTIONS:
Other: Understanding Needs Survey — 2-hour Focus Group
  Mailed or E-mailed Survey

SUMMARY:
The "Understanding Needs" Project is designed to gain an understanding of the needs of informal caregivers. Researchers have designed a survey to highlight activities of daily living involved in the caregiving role, pain related to caregiver, and potential services desired. The initial phase of the study will consist of a focus group of informal caregivers to discuss current needs. The survey will then be refined based on knowledge gained from the focus group, and feedback from expert researchers. The refined survey will then be disseminated to caregivers throughout the country.

Please click on the following anonymous link to participate: https://chhscolostate.co1.qualtrics.com/jfe/form/SV_54j83BQSItMuoUB

DETAILED DESCRIPTION:
The "Understanding Needs" Project highlights the needs of informal caregivers. An informal caregiver is defined as a person who regularly provides unpaid care to another adult. The survey will ask about pain intensity, pain interference, and relation of pain to the caregiving role. The survey will also address which activities the caregiver assists with, and activities now lacking since becoming a caregiver. One focus group will be completed to refine the contents of the survey prior to dissemination. The results will be analyzed by an occupational therapist, with a focus on how pain may connect to assistance with daily living activities provided to the care recipient. The needs of caregivers within the community will be compiled to inform future involvement in remediation of needs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Informal caregivers (unpaid)
* have been a caregiver for > 6 months
* provide at least 8 hours of care/week
* able to read english

Exclusion Criteria:

* Less than 18 years old
* paid caregivers
* not able to read english
* Caregiver or care recipient has a terminal diagnosis with a life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
PEG: Three Item Pain Measure | Self-report, up to one year for analyses when all surveys are returned
  A self-rating of pain intensity, pain interference in enjoyment of life, and pain interference in general activity

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No